CLINICAL TRIAL: NCT06370871
Title: Brightline-3: A Phase III, Randomized, Open-label, Multi-center Trial of Brigimadlin + Ezabenlimab Compared to Gemcitabine + Docetaxel for Second-line Treatment of Patients With Advanced TP53 Wild-type Soft Tissue Sarcoma Subtypes
Brief Title: Brightline-3: A Study to Find Out Whether Brigimadlin in Combination With Ezabenlimab Helps People With Advanced Soft Tissue Sarcoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0006; 2022-502985-26-00 (Registry Identifier: CTIS (EU)); U1111-1292-9594 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Advanced Soft Tissue Sarcoma; Undifferentiated Pleomorphic Sarcoma (UPS); Myxofibrosarcoma (MFS)
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma | interventions — brigimadlin; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Ezabenlimab (Experimental)
  Interventions: Drug: Ezabenlimab
- Arm B: Brigimadlin + ezabenlimab (Experimental)
  Interventions: Drug: Brigimadlin; Drug: Ezabenlimab
- Arm C: Gemcitabine + docetaxel (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Brigimadlin — Brigimadlin
  Other Names: BI 907828
  Arms: Arm B: Brigimadlin + ezabenlimab
Drug: Ezabenlimab — Ezabenlimab
  Other Names: BI 754091
  Arms: Arm A: Ezabenlimab; Arm B: Brigimadlin + ezabenlimab
Drug: Gemcitabine — Solution for infusion
  Arms: Arm C: Gemcitabine + docetaxel
Drug: Docetaxel — Solution for infusion
  Arms: Arm C: Gemcitabine + docetaxel

SUMMARY:
This study is open to adults with specific types of advanced soft tissue sarcoma. People with undifferentiated pleomorphic sarcoma (UPS) or myxofibrosarcoma (MFS) can join the study if they have a normal version of the TP53 gene. This is a study for people whose earlier treatment isn't working anymore, and their doctors suggest a new treatment to stop the sarcoma from getting worse.

The purpose of this study is to compare a medicine called brigimadlin in combination with another medicine called ezabenlimab with chemotherapy. Brigimadlin is a so-called MDM2-p53 antagonist that is being developed to treat cancer. Ezabenlimab is an antibody that may help the immune system fight cancer.

Participants are put into 3 groups by chance:

* Ezabenlimab group: Participants receive ezabenlimab as an infusion into a vein every 3 weeks
* Brigimadlin + ezabenlimab group: Participants take brigimadlin as tablets and receive ezabenlimab as an infusion into a vein every 3 weeks
* Chemotherapy group: Participants get chemotherapy as an infusion into a vein on 2 days every 3 weeks. Chemotherapy is a combination of gemcitabine and docetaxel which is often used in the treatment of sarcoma.

There are twice as many participants in the brigimadlin + ezabenlimab group and in the chemotherapy group, compared to those in the ezabenlimab group.

Participants can continue treatment in the study as long as they benefit from it and can tolerate it.

Doctors regularly check the size of the tumor and check whether it has spread to other parts of the body. The doctors also regularly check participants' health and take note of any unwanted effects. Participants in this study use an app on a mobile phone to regularly answer questions about their health and well-being. This is to find out if their quality of life is changing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form (ICF) in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good clinical practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses
2. Male or female patients ≥18 years old at the time of signature of the ICF
3. Histologically proven diagnosis of one of the following:

   * Undifferentiated pleomorphic sarcoma (UPS) with TP53 wild-type status
   * Myxofibrosarcoma (MFS) with TP53 wild-type status
4. Written pathology report indicating the diagnosis of UPS or MFS must be available
5. Written report from the trial central laboratory indicating TP53 wild-type status
6. One prior systemic regimen for advanced disease with documented progressive disease as per serial radiologic imaging. If prior systemic cytotoxic treatment for soft tissue sarcoma was given in a neoadjuvant, adjuvant or perioperative setting that treatment would count as one line of therapy in case of radiological progression during that treatment or within 3 months after completing that systemic therapy. If progression or relapse occurred after >3 months after completing that systemic therapy, the pre-, post or perioperative treatment would not count as a line of treatment for advanced disease
7. Patient must be willing to donate mandatory blood and tissue samples for the pharmacokinetics, pharmacodynamics, and biomarker analyses
8. Presence of at least one target lesion according to RECIST Version 1.1 Further inclusion criteria apply

Exclusion Criteria:

1. Prior treatment with immunotherapy in the context of anticancer therapy
2. Previous administration of gemcitabine, taxanes, brigimadlin or any other mouse double minute 2 homolog-p53 (MDM2-p53) or MDMX (MDM4)-p53 antagonist
3. Previous or concomitant malignancies other than the one treated in this trial within the previous 2 years, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or other malignancy that is considered cured by local treatment
4. Patient unable to swallow the trial medication
5. Any history or presence of uncontrolled gastrointestinal disorders that could affect the intake and/or absorption of the trial drug (e.g., nausea, vomiting, Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption) in the opinion of the investigator
6. Active bleeding, significant risk of hemorrhage (e.g., previous severe gastrointestinal bleeding, previous hemorrhagic stroke at any time), or current bleeding disorder (e.g., hemophilia, von Willebrand disease)
7. Known history of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity or known contraindication to the trial medications or their excipients
8. Active autoimmune disease or a documented history of autoimmune disease, that requires systemic treatment, i.e., corticosteroids or immunosuppressive drugs, except for vitiligo or resolved childhood asthma/atopy, alopecia, or any chronic skin condition that does not require systemic therapy; patients with autoimmune-related hypothyroidism on a stable dose of thyroid hormone replacement and/or controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-27 (Estimated); Primary Completion 2026-07-03 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 4 years.
  Progression-free survival is defined as the time from randomization until the earliest of tumor progression according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1, based on blinded central independent review or death from any cause.
Overall survival | up to 4 years.
  Overall survival, defined as the time from randomization until death from any cause.

SECONDARY OUTCOMES:
Objective response | up to 4 years.
  Objective response (OR), defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST Version 1.1 (based on central independent review) from the date of randomization until the earliest of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Duration of objective response | up to 4 years.
  Duration of objective response (DOR), defined as the time from first documented confirmed OR according to RECIST Version 1.1 until the earliest of disease progression or death among patients with confirmed objective response (based on central independent review).
Disease control | up to 4 years.
  Disease control (DC), defined as a best overall response of CR, PR, or stable disease (SD), where best overall response is defined according to RECIST Version 1.1 (based on central independent review).
Duration of disease control | up to 4 years.
  Duration of disease control, defined as the time from randomization until the earliest of disease progression according to RECIST Version 1.1 (based on central independent review) or death from any cause among patients with disease control.
Occurrence of treatment-emergent adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5 | up to 4 years.
Occurrence of treatment-emergent AEs leading to study drug discontinuation | up to 4 years.
Mean change from baseline to Week 12 in the domain fatigue (based on items from the European Organization for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) and the EORTC item library) | At baseline and at Week 12.
  Fatigue will be assessed via 8 items. The score of each item ranges from 0-100 with higher scores indicating higher symptomology.
Mean change from baseline to Week 12 in the domain fatigability (based on items from the EORTC QLQ-C30 and the EORTC item library) | At baseline and at Week 12.
  Fatigability will be assessed via 12 items. The score of each item ranges from 0-100 with higher scores indicating higher symptomology.
Mean change from baseline to week 12 in the domain physical functioning (based on items from the EORTC QLQ-C30) | At baseline and at Week 12.
  EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes (PROs). The gloabl health status and the quality of life are 2 of the 30 items and are scored from 1 (1=very poor) to 7 (7=excellent).
  All other items have 4 possible scores (1= not at all, 2= a little, 3=quite a bit, 4=very much).
Mean change from baseline to week 12 in the domain pain (based on items from the EORTC QLQ-C30) | At baseline and at Week 12.
  EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes (PROs). The gloabl health status and the quality of life are 2 of the 30 items and are scored from 1 (1=very poor) to 7 (7=excellent).
  All other items have 4 possible scores (1= not at all, 2= a little, 3=quite a bit, 4=very much).
Mean change from baseline to week 12 in the domain dyspnea (based on items from the EORTC QLQ-C30) | At baseline and at Week 12.
  EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes (PROs). The gloabl health status and the quality of life are 2 of the 30 items and are scored from 1 (1=very poor) to 7 (7=excellent).
  All other items have 4 possible scores (1= not at all, 2= a little, 3=quite a bit, 4=very much).
Mean change from baseline to week 12 in the domain global health status / quality of life (based on items from the EORTC QLQ-C30) | At baseline and at Week 12.
  EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes (PROs). The gloabl health status and the quality of life are 2 of the 30 items and are scored from 1 (1=very poor) to 7 (7=excellent).
  All other items have 4 possible scores (1= not at all, 2= a little, 3=quite a bit, 4=very much).

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com